CLINICAL TRIAL: NCT02244970
Title: Brief Mindfulness-Based Intervention for Early Psychosis: A Randomized Controlled Study
Brief Title: Mindfulness RCT for Early Psychosis
Acronym: MBIp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Eric Y H Chen, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIND2014
Record Dates: First submitted 2014-08-21; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Psychosis
Keywords: Mindfulness; Depressive mood; anxiety; early psychosis
MeSH Terms: conditions — Psychotic Disorders; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness (Experimental): Subjects are scheduled to receive a 7-week group mindfulness-based intervention (MBI) program.
  Interventions: Other: Mindfulness
- Psychoeducation (Active Comparator): Subjects will receive 7 weeks of group-based psychoeducation as an active comparison group parallel to the mindfulness group.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: Mindfulness — Mindfulness is the awareness that emerges from paying attention to the present moment without judgment. In this study, subject in this arm will receive 7 weeks of MBI with a focus on tackling anxiety, depressed mood, and attention deficits among early psychosis participants. The elements of 7-week program included mindful-breathing, indoor and outdoor mindful-walking, mindful-eating, mindul-drawing, tree-of-life exercise and closing celebration.
  Arms: Mindfulness
Other: Psychoeducation — Participants in the psychoeducation group will receive seven weeks of psychoeducation sessions which include basic knowledge related to 1) General mental health, 2) Knowledge of psychosis, 3) Treatment and community resources, 4) Recovery and relapse prevention, 5) Healthy lifestyle, 6) Social skills training, and finally a closing celebration at week 7.
  Arms: Psychoeducation

SUMMARY:
Depressive mood and anxiety are prevalent in patients suffering from early psychosis. Treatments focused on these dimensions are rarely seen. Meanwhile, growing evidence showed Mindfulness-based intervention (MBI) as an effective option in handling depression and anxiety. There is a great possibility that MBI is also useful in depression and anxiety associating with early psychosis. Given that cost-effectiveness is widely concerned in Hong Kong or any other countries, a brief intervention is more favored. Current paper is a study protocol for a randomized controlled trial which assess the feasibility of a 7-week mindfulness-based intervention in patients with early psychosis targeting on their depressive mood and anxiety.

In this RCT, 60 patients aged 18-65 with early psychosis less than 5 years' duration and mild depressive mood or anxiety will be invited to join this single blind randomized controlled trial. After baseline assessments, eligible participants will be, using third party simple randomization, randomly assigned to either the 7-week Mindfulness-based Intervention (MBI), or the psychoeducation group as control.

The primary outcome is depressive mood and anxiety levels at post-intervention and 3 months. The secondary outcomes include life functioning, quality of life, other general clinical symptoms and mindfulness ability. Qualitative interviews will help evaluate and measure the feasibility of the intervention. Data will be analyzed according to the intention-to-treat principle.

This randomized trial offers an insight into mindfulness-based intervention and its effectiveness on psychosis concomitants. It provides the foundation for future evaluation and implementation of an effective and cost-efficient treatment option.

DETAILED DESCRIPTION:
Psychosis is a set of symptoms associated with distorted perception and cognition. Clinical treatments that focus on positive symptoms, hallucination, and delusion are increasingly well developed throughout the century. However peripheral facets such as depressive mood (post-psychotic depression to its extreme) and anxiety have never been the foci of attention; they are often viewed as less important than positive, negative, or cognitive symptoms, if not entirely ignored. Sadly, depression and anxiety are prevalent in early psychotic patients. Depression was found in 22% of people with First Episode Psychosis (FEP), and anxiety disorders of social phobia was found in 32%, and obsessive compulsive disorder in 4-15% of people with FEP. These adverse conditions after the early acute stage of psychosis are linked with poor engagement in treatment services and adverse impact on the change process, resulting in poor treatment outcomes, lowered quality of life, and increased likelihood of suicide. Given the high prevalence and extensive impact, there is a need to explore adjunction intervention that targets mood and anxiety symptoms following onset of psychotic disorders.

Mindfulness is the awareness that emerges from paying attention to the present moment without judgment. It is a skill that can be achieved through meditation practices, and has been shown to improve general well-being. Mindfulness-based intervention (MBI) has been referred to as the "third wave" of psychological interventions after the first wave behavioral and the second wave cognitive interventions. Research relating to MBIs has increased exponentially in the past decade. Key, fully developed, MBIs in the literature include mindfulness-based stress reduction (MBSR), mindfulness-based cognitive therapy (MBCT) and acceptance and commitment therapy (ACT). These interventions are increasingly used with individuals suffering from depression or anxiety and have gained positive findings. Hofmann and colleagues conducted an effect size analysis on 39 studies of MBI for anxiety and mood symptoms in clinical samples. They found a moderately strong uncontrolled pre-post effect size of MBIs on reducing anxiety symptoms and depressive symptoms among individuals with disorders not limited to anxiety disorders or major depression. The authors postulated that MBIs may not be diagnosis-specific. Rather it is effective in reducing stress in general and hence improves symptoms of anxiety and depression across a relatively wide range of conditions.

Since MBIs are efficacious in reducing mood and anxiety symptoms across various disorders, it has potential intervention value for early psychosis as well. In a recent meta-review, Khoury and colleagues concluded that MBIs have moderate therapeutic effects for psychosis. At the same time, there are arguments against mindfulness practices on active psychotic patients, and in people at risk of developing psychosis. In response, Chadwick et al. demonstrated in a feasibility study the safe use of a mindfulness intervention on nine active psychotic patients. Given the small sample size, further careful research, especially randomized controlled trials (RCTs), is needed to support its usage .

Evidence on mindfulness-based interventions in treatment of mood and anxiety symptoms is encouraging. Yet, only a small number of RCTs have been conducted on patients with early psychosis to date. Further, with the limited resources available to the health system in Hong Kong, we aimed to create a simple MBI specific for early psychosis patients, with a user-friendly protocol that can be operated by health practitioners after sufficient yet time-efficient training. Therefore, the current RCT protocol in assessing the efficacy of a brief MBI on patients with early psychosis is of value.

The primary research question is whether positive changes on depressive and anxiety symptoms can be obtained through a 7-week MBI program designed for early psychotic patients. Specifically, we hypothesized that the anxiety level and depressive mood can be significantly reduced by our MBI. The second question we sought to answer is whether this change can be maintained, as reflected in a 3-month follow up. Our secondary hypotheses are that since depression and anxiety are lowered, those receiving the MBI will perceive having better quality of life and overall functioning as a result

ELIGIBILITY:
Inclusion Criteria:

* Cantonese-speaking patients aged 18-65, who are service users of the aforementioned community mental health services in Hong Kong.
* diagnosis of Schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, psychotic disorder not otherwise specified, or manic episodes with psychotic features according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) and less than 5 years' duration since onset of psychosis.
* present with mild depressive or anxiety symptoms (PANSS items G2 or G6 scores higher than or equal to 3; any item on CDSS scores more than or equal to 1).
* They must have an ability to consent, stable positive symptoms (PANSS symptomatic items: P1-P7 scores less than or equal to 3) and good medication compliance (assessed by clinical interview, informant interview, and pill-counting).

Exclusion Criteria:

* Known organic brain disorder
* Known history of intellectual disability,
* Diagnosed with drug-induced psychosis,
* Practice of mindfulness (in forms of yoga, Tai Chi, etc.) more than twice a week during the previous three months,
* Previous or current substance abuse,
* High risk features associated with acute psychotic episodes, and
* Questionable adherence to medication treatment and follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Depressive mood | 19weeks
  Depressive mood is measured by the Positive and Negative Symptom Scale Item G2 (PANSS-G2); Calgary Depression Scale for Schizophrenics (CDSS); Depression Anxiety Stress Scale - Depression subscale (DASS-21-D) and Beck Depression Inventory - II (BDI-II).
Anxiety | 19weeks
  Anxiety is measured by DASS-21 - Anxiety subscale and PANSS item G6.

SECONDARY OUTCOMES:
Quality of Life | 19weeks
  measured by Short Form 12 (SF12)
Life Functioning | 19weeks
  rated on the Social and Occupational Functioning Assessment Scale (SOFAS)
Mindfulness | 19weeks
  two separate mindfulness scales: the Five Facet Mindfulness Questionnaire (FFMQ) and the Southampton Mindfulness Questionnaire (SMQ).We also take note of the number of practices conducted individually by participants during each week of the intervention period and also the frequency of practice after the seven weeks of MBI.

OTHER OUTCOMES:
Program evaluation | 19weeks
  In order to evaluate the MBI for further development and to assist interpretation of results, qualitative semi-structured interviews will be conducted after the seven weeks of MBI. The interview primarily looks at the perceived processes of change, helpful aspects of the process, and therapeutic value of the MBI. Each interview will be recorded and transcribed

CONTACTS AND LOCATIONS:
Overall Officials: JingXia Lin, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China